CLINICAL TRIAL: NCT05229640
Title: Relationship Between the Development of Impaired Glucose Tolerance, the Phenotype of CFLD, and the Risk of Liver Fibrosis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Trustees of Dartmouth College (Other)
Responsible Party: Principal Investigator, Mary C. Drinane, Principal Investigator, Staff Physician, Gastroenterology & Hepatology, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY02001342
Record Dates: First submitted 2021-12-21; First posted 2022-02-08 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: CF - Cystic Fibrosis; Cystic Fibrosis-related Diabetes; Cystic Fibrosis Liver Disease
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Fibroscan (Other): One study visit for fibroscan measurement of the liver.
  Interventions: Device: Fibroscan

INTERVENTIONS:
Device: Fibroscan — Subjects will fast for at least three hours, then have at least 10 fibroscan readings of their liver.

SUMMARY:
This study proposes to examine the relationship between the development of impaired glucose tolerance, the phenotype of CFLD, and risk of liver fibrosis.

DETAILED DESCRIPTION:
Pancreas insufficiency is a well-established risk factor for development of CF related diabetes (CFRD), but increased insulin resistance has also been demonstrated in this population. Cystic fibrosis liver disease (CFLD) is a well-established risk factor for the development CFRD. In addition, patients with CFLD and CFRD at high risk of development of severe CFLD and cirrhosis. Recent work has shown that male CF patients with abnormal oral glucose tolerance tests were noted to have elevations in ALT but the significance of this finding has yet to be fully explored. Specifically, an unresolved question remains on whether the elevation in ALT reflects a steatohepatitis as would be observed in a non-CF population or if the increased insulin resistance contributes to fibrosis progression in the classic biliary type cirrhosis seen in cystic fibrosis (CF).

Metabolic dysfunction with increasing insulin resistance has been shown to be a key component to the development of non-alcoholic steatosis hepatitis in a non-CF population. The presence of hepatic steatosis has been demonstrated in the CF population, but thus far not been linked to the development of significant steatohepatitis or cirrhosis. One potential explanation for this discordance between effects of hepatic steatosis in the CF and non-CF population, is in the non-CF population it requires multiple decades for hepatic steatosis to result in steatohepatitis and progression to cirrhosis, therefore the progressive fibrosis may not be seen in the CF population due to limited life expectancy. However, as the life expectancy in of patients with CF is increasing with new therapy, the longer-term consequences of hepatic steatosis maybe apparent

Alternatively, the presence of increased insulin resistance has been correlated to increase fibrosis progression in other forms of liver disease such as hepatitis C. Therefore, another potential mechanism is the insulin resistance seen in patients with CFRD results in increased fibrosis and development of cirrhosis in patients with classic CFLD. Thus, further characterizing the underlying liver disease phenotype and fibrosis risk in this population is of interest. We propose to examine the relationship between the development of impaired glucose tolerance, the phenotype of CFLD, and risk of liver fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 with CF and one of the following:

  * Normal OGTT
  * Elevated OGTT
  * Known CFRD

Exclusion Criteria:

* Men and women without CF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Assess Phenotype of CFLD | Visit 1, Day 1
  Assess phenotype of CFLD via a Fibroscan performed after a >3 hour fast
Assess Value of Complete Blood Count of CFLD | Visit 1, Day 1
  Assess phenotype of CFLD via a complete blood count (CBC)
Assess Hepatic Function of CFLD | Visit 1, Day 1
  Assess phenotype of CFLD via a hepatic function test
Assess Oral Glucose of CFLD | Visit 1, Day 1
  Assess phenotype of CFLD via an oral glucose tolerance test
Assess CFLD via abdominal imaging | Visit 1, Day 1
  Assess phenotype of CFLD via abdominal imaging (CT abdomen, Ultrasound, or MRI). If the subject has had a CT of the abdomen, Ultrasound or MRI of the abdomen as part of their standard care, the data will be collected. These procedures will not be performed as part of this study.

CONTACTS AND LOCATIONS:
Overall Officials: Mary C. Drinane, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available to other researchers.

REFERENCES:
- [Result] Kayani K, Mohammed R, Mohiaddin H. Cystic Fibrosis-Related Diabetes. Front Endocrinol (Lausanne). 2018 Feb 20;9:20. doi: 10.3389/fendo.2018.00020. eCollection 2018. PMID 29515516
- [Result] Toledano MB, Mukherjee SK, Howell J, Westaby D, Khan SA, Bilton D, Simmonds NJ. The emerging burden of liver disease in cystic fibrosis patients: A UK nationwide study. PLoS One. 2019 Apr 4;14(4):e0212779. doi: 10.1371/journal.pone.0212779. eCollection 2019. PMID 30947265
- [Result] Colomba J, Netedu SR, Lehoux-Dubois C, Coriati A, Boudreau V, Tremblay F, Cusi K, Rabasa-Lhoret R, Leey JA. Hepatic enzyme ALT as a marker of glucose abnormality in men with cystic fibrosis. PLoS One. 2019 Jul 18;14(7):e0219855. doi: 10.1371/journal.pone.0219855. eCollection 2019. PMID 31318914
- [Result] Friedman SL, Neuschwander-Tetri BA, Rinella M, Sanyal AJ. Mechanisms of NAFLD development and therapeutic strategies. Nat Med. 2018 Jul;24(7):908-922. doi: 10.1038/s41591-018-0104-9. Epub 2018 Jul 2. PMID 29967350
- [Result] Hui JM, Sud A, Farrell GC, Bandara P, Byth K, Kench JG, McCaughan GW, George J. Insulin resistance is associated with chronic hepatitis C virus infection and fibrosis progression [corrected]. Gastroenterology. 2003 Dec;125(6):1695-704. doi: 10.1053/j.gastro.2003.08.032. PMID 14724822